CLINICAL TRIAL: NCT01162863
Title: A Pilot Study to Assess the Effects of Lubiprostone on Gastrointestinal and Colonic Motility and pH in Patients With the Irritable Bowel Syndrome and Constipation (IBS-C)
Brief Title: Effects of Lubiprostone on Gastrointestinal Transit & pH in Irritable Bowel Syndrome (IBS) With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Richard J. Saad, M.D., Assistant Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 08-028LUB
Record Dates: First submitted 2010-07-09; First posted 2010-07-15 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Irritable Bowel Syndrome; Constipation
Keywords: IBSC; irritable bowel syndrome; constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Lubiprostone 8 mcg BID (Active Comparator)
  Interventions: Drug: Lubiprostone; Other: Smartpill wireless motility capsule
- Lubiprostone 24 mcg QD (Active Comparator)
  Interventions: Drug: Lubiprostone; Other: Smartpill wireless motility capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Smartpill wireless motility capsule

INTERVENTIONS:
Drug: Lubiprostone — lubiprostone taken either at a dose of 8 mcg orally twice daily (BID) for 28 days or 24 mcg orally once daily (QD) for 28 days
  Arms: Lubiprostone 24 mcg QD; Lubiprostone 8 mcg BID
Drug: Placebo — taken orally for 28 days
  Arms: Placebo
Other: Smartpill wireless motility capsule — Ingestion of a small non-digestible capsule that measures temperature, pH and pressure of the immediate surrounds as it passes through the GI tract eventually exiting the body through the anus

SUMMARY:
Irritable bowel syndrome (IBS) is a common disorder which presents with abdominal pain or discomfort in association with altered bowel habit. IBS is further subcategorized as three types according to the predominant bowel movement pattern: IBS with constipation (IBS-C), IBS with diarrhea (IBS-D), and mixed-IBS (IBS-M). The exact causes of IBS remain incompletely understood, but proposed mechanisms include abnormal motility, visceral hypersensitivity, abnormal brain-gut interactions, psychological distress, and altered GI tract motility.

Lubiprostone, a novel drug that works by activating the colonic Chloride channel type 2(ClC-2), has been approved for use in patients with chronic idiopathic constipation and recently approved for the treatment of IBS-C in women aged 18 and older. By activating the ClC-2 chloride channel in the colon, lubiprostone allows more fluid secretion into the intestinal lumen which leads to softer stool consistency. In phase III clinical trials, patients with IBS-C receiving lubiprostone have reported improvements in many symptoms such as abdominal pain and constipation. However, there is limited physiologic data to explain how exactly lubiprostone improves IBS-C symptoms.

The Smartpill is a novel non-digestible capsule that is capable of measuring intraluminal pH, pressure, and temperature in the gastrointestinal (GI) tract. Smartpill has been shown to accurately measure whole gut as well as regional (i.e. stomach, small bowel, colon) transit time.

The primary aim of this study is to determine the effects of lubiprostone on whole GI tract transit, colonic transit, motility, and intraluminal pH in patients with IBS-C through evaluation with the Smartpill. The investigators propose to study the effect of lubiprostone vs. placebo on these parameters, and secondarily to evaluate changes in these parameters with differing doses of lubiprostone.

The investigators hypothesize that lubiprostone will increase whole GI and colonic transit compared to placebo in patient with IBS. the investigators do not expect a change in intraluminal pH with lubiprostone compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females >18 years of age
* Meet Rome III criteria for IBS[2]:

  * Recurrent abdominal pain or discomfort at least 3 days per month in the last 3 months associated with 2 or more of the following:

    1. Improvement with defecation
    2. Onset associated with a change in frequency
    3. Onset associated with a change in form (appearance) of stool
  * *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
* Fulfill the Rome III stool consistency criteria for IBS-C[2]

  * Hard or lumpy stools for >25% of bowel movements
  * Loose (mushy) or watery stools for <25% of bowel movements
* Capable of independently completing all requirements of the study including returning for required visits
* Able to provide written informed consent for study participation
* Willing to discontinue prohibited medications during study participation
* Documentation of a normal colonoscopy within last 5 years if over age 50 years (or sigmoidoscopy if less than age 50)
* Documentation of normal thyroid stimulating hormone(TSH) level, complet blood count (CBC) and electrolyte panel within prior 3 years
* Females of childbearing potential must have a negative urine or serum pregnancy test at screening
* Females of childbearing potential must use an effective means of contraception during the course of the study

  * Hormonal (oral, injectable, implantable, cervical/vaginal rings or patches)
  * Double-barrier (condoms and/or diaphragm with spermicides) or intrauterine devices provided under the care of a health care professional
  * Abstinence, in this case documentation of counseling will be recorded

Exclusion Criteria:

* Unable to understand or provide written informed consent
* Pregnant or nursing
* Patients with IBS-D, IBS-M or unsubtyped IBS by Rome III criteria[2]
* IBS with diarrhea (IBS-D)

  1. Loose (mushy) or watery stools for >25% of bowel movements
  2. Hard or lumpy stools for <25% of bowel movements
* Mixed IBS (IBS-M)

  1. Hard or lumpy stools >25% of bowel movements
  2. Loose (mushy) or watery stools for >25% of bowel movements
* Unsubtyped IBS

  1. Insufficient abnormality of stool pattern to meet criteria for IBS-C, IBS-D or IBS-M
* Documented allergy or intolerance to lubiprostone
* Failure of balloon expulsion test

  * Inability to expel 50cc balloon within 1 minute
* Use of drugs known to affect gastrointestinal motility

  1. Laxatives (stable doses of fiber taken for minimum of 4 weeks will be allowed)

     Osmotic laxatives:

     Magnesium hydroxide, Polyethylene glycol,Lactulose, Sorbitol

     Stimulant laxatives:

     Bisacodyl, Anthraquinones (senna), Misoprostol
  2. Prokinetic agents:

     Metoclopramide, domperidone, erythromycin
  3. Anti-diarrheal agents:

     Loperamide, Diphenoxylate, Bismuth
  4. Anti-spasmotics:

     Dicyclomine, Hyoscyamine
  5. Opioid, narcotic, opioid/narcotic-containing analgesics:

     Morphine, Hydrocodone, Codeine, Methadone, Propoxyphene
  6. Probiotics
  7. Systemic antibiotics within last 3 months
  8. Recently initiated antidepressants (stable dose for >2 months for non-GI conditions will be allowed)
  9. Benzodiazepines * Subjects taking prohibited medications will be required to stop these at the screening visit and remain off of them until completion of the study.
* Initiation of dietary changes potentially altering bowel transit within 4 weeks
* Comorbid medical problems that may affect gastrointestinal transit or motility

  1. Previous surgery involving the stomach, small bowel or colon (prior appendectomy, cholecystectomy, polypectomy allowed)
  2. Previous history of small bowel obstruction for any reason
  3. History of any gastrointestinal malignancy
  4. History of dyssynergic defecation
  5. Unexplained nausea and vomiting
  6. History of inflammatory bowel disease (Crohn's or ulcerative colitis)
  7. History of microscopic colitis (lymphocytic or collagenous colitis)
  8. History of Hirschsprung's disease
  9. Severe or complicated diverticular disease
  10. Chronic pancreatitis
  11. History of celiac disease
  12. History of eating disorders (anorexia nervosa or bulimia)
  13. Cirrhosis
  14. Chronic hepatitis B or C infection
  15. HIV infection
  16. Diabetes
  17. Systemic sclerosis (scleroderma)
  18. Amyloidosis
  19. Untreated thyroid disease
  20. Chronic pulmonary disease
  21. Severe renal insufficiency or renal failure
  22. Current or recent history (within last 6 months) of:

      Diverticulitis, Duodenal or gastric ulcer, Acute pancreatitis, Ileus
* Contraindications to SmartPill® (in addition to above):

Cardiac pacemaker, defibrillator, or other implanted electromagnetic device, Known Zenker's diverticulum, Dysphagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saad, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 adults were screened of whom 4 were screen failures.Of the 56 remaining study participants, 2 were unable to swallow the wireless motility capsule and 2 more dropped out of the study prior to randomization yielding 52 randomized participants.
Groups:
- Lubiprostone 24 mcg QD; Lubiprostone 8 mcg BID: Lubiprostone: lubiprostone taken either at a dose of 8 mcg orally twice daily for 28 days or 24 mcg orally once daily for 28 days
  Smartpill wireless motility capsule: Ingestion of a small non-digestible capsule that measures temperature, pH and pressure of the immediate surrounds as it passes through the GI tract eventually exiting the body through the anus
Period: Overall Study
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID
Started | 18 | 17 | 17
Completed | 17 | 16 | 17
Not Completed | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline data is given for those persons who actually completed the study, so the two people who dropped out were not included in the baseline measures. We determined this to be the more useful way to identify the effects of the three randomized procedures. Therefore the baseline data is based on the 50 participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID | Total
Number analyzed (Participants) | 17 | 16 | 17 | 50
Age, Customized [Mean (Standard Deviation); unit: years]
  mean age | 39.9 (16.1) | 46.5 (18.7) | 37.2 (15.8) | 41.2 (17.2)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 15 | 13 | 44
  Male | 1 | 1 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 17 | 50
Baseline gastric emptying time [Mean (Standard Deviation); unit: hours] | 4.25 (5.52) | 3.18 (0.95) | 4.67 (3.47) | 4.01 (3.74)
Baseline Small Bowel Transit time [Mean (Standard Deviation); unit: hours] | 4.84 (1.69) | 4.01 (1.02) | 4.81 (2.13) | 4.63 (1.75)
Baseline Colon Transit Time [Mean (Standard Deviation); unit: hours] | 32.18 (16.46) | 44.61 (27.18) | 37.12 (30.04) | 38.15 (25.31)
Baseline Whole Gut Transit Time [Mean (Standard Deviation); unit: hours] | 41.47 (16.26) | 51.81 (26.78) | 47.0 (30.0) | 47.0 (24.97)
Baseline Small Bowel pH [Mean (Standard Deviation); unit: units on pH scale] | 6.82 (0.28) | 6.75 (0.34) | 6.77 (0.39) | 6.78 (0.33)
Baseline Colon pH [Mean (Standard Deviation); unit: units on pH scale] | 6.56 (0.55) | 6.75 (0.34) | 6.47 (0.48) | 6.50 (0.51)
Baseline Small Bowel Motility Index [Mean (Standard Deviation); unit: units on a scale] — natural log [(sum of pressure amplitudes times the number of contractions) + 1] , resulting in a sort of units on a naturally derived scale
  units on a scale | 13.14 (1.66) | 12.80 (1.86) | 12.65 (2.26) | 12.86 (1.93)
Baseline Colon Motility Index [Mean (Standard Deviation); unit: units on a scale] — natural log [(sum of pressure amplitudes times the number of contractions) + 1]
  units on a scale | 16.26 (1.57) | 16.9 (2.14) | 16.17 (1.79) | 16.43 (1.83)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastric Emptying Time, Small Bowel Transit Time, Colon Transit Time and Whole Gut Transit Time From Baseline
Description: Change in gastric emptying time, small bowel transit time, colon transit time and whole gut transit time measured in hours based on a measurement done at baseline and then again at 3 weeks into the intervention within each treatment arm
Time Frame: 21-28 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID
Number analyzed (Participants) | 17 | 16 | 17
hours
  Gastric emptying time | 5.49 (13.77) | 6.52 (15.33) | -0.16 (3.17)
  Small bowel transit time | 0.2 (2.04) | 0.15 (1.78) | -0.001 (2.68)
  Colon transit time | 5.75 (21.23) | -4.43 (44.6) | 2.59 (31.15)
  Whole gut transit time | 10.32 (27.3) | -1.74 (42.67) | 1.67 (29.73)

2. Secondary Outcome: Change in Small Bowel pH and Colon pH From Baseline
Description: Change in the mean pH of the small intestine and colon based on a measurement done at baseline and then again at 3 weeks into the intervention.
Time Frame: 21-28 days
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID
Number analyzed (Participants) | 17 | 16 | 17
pH
  Small bowel pH | 0.18 (0.37) | 0.23 (0.36) | 0.24 (0.4)
  Colon pH | -0.03 (0.50) | -0.07 (0.45) | 0.27 (0.56)

3. Secondary Outcome: Change in Motility Pattern of the Small Bowel and Colon From Baseline as Defined by the Motility Index
Description: Change in the motility index defined as the natural log [(sum of pressure amplitudes times the number of contractions) + 1] for the small bowel and colon based on a measurement done at baseline and then again at 3 weeks into the intervention.
Time Frame: 21-28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID
Number analyzed (Participants) | 17 | 16 | 17
units on a scale
  Small bowel motility index | 0.06 (1.37) | -0.01 (1.89) | 0.6 (2.36)
  Colon motility index | -0.34 (1.96) | -1.32 (1.97) | 0.17 (1.72)

ADVERSE EVENTS:
Arm/Group | Placebo | Lubiprostone 24 mcg QD | Lubiprostone 8 mcg BID
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 9/18 | 11/17 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Lubiprostone 24 mcg QD (N=17) | Lubiprostone 8 mcg BID (N=17)
Dehydration (Cardiac disorders) | 1 | 0 | 0 — brief hospitalization for dehydration and disorientation at end of treatment phase
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 — Episode of atrial fibrillation spontaneously resolving
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=18) | Lubiprostone 24 mcg QD (N=17) | Lubiprostone 8 mcg BID (N=17)
Diarrhea (Gastrointestinal disorders) | 2 | 6 | 4/16
Nausea (Gastrointestinal disorders) | 4 | 6 | 6
Headache (General disorders) | 1 | 2 | 2
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 4 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 2
Abdominal distention (Gastrointestinal disorders) | 0 | 2 | 4
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
This was a small study with wide variability among participants, so data should be interpreted with great caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No